CLINICAL TRIAL: NCT04837885
Title: "Imaging With 68Ga-DOTA-peptides and Peptide Receptor Radionuclide Therapy With 177Lu-DOTA-peptides of Gastroenteropancreatic Neuroendocrine Tumors: Interest of Intra-arterial Hepatic Infusion in Patients With Dominant Liver Metastases"
Brief Title: Intra-arterial Hepatic (IAH) Infusion of Radiolabelled Somatostatin Analogs in GEP-NET Patients With Dominant Liver Metastases
Acronym: LUTARTERIAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2017/47
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neuroendocrine Tumor; Liver Metastases; Neuroendocrine Gastroenteropancreatic Tumour
Keywords: Neuroendocrine tumour; Neuroendocrine gastroenteropancreatic (GEP) tumour; Liver Metastases; 68Ga- DOTA-peptides PET CT; 177Lutetium-Octreotate; Peptide Receptor Radionuclide Therapy
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-peptides PET/CT (Experimental): 68Ga-DOTA-peptides injections for targeted liver metastases in Positron emission tomography-computed tomography (PET/CT)
  One treatment dose of LUTATHERA® by intra-arterial hepatic injection (IAH) after conventional treatment by 4 intravenous administrations
  Interventions: Procedure: Positron emission tomography computed tomography (PET/CT) with Intra-hepatic (IAH) injection; Procedure: Positron emission tomography computed tomography (PET/CT) with Intravenous (IV) injection; Drug: LUTATHERA® by intra-arterial hepatic (IAH) injection; Procedure: Scan

INTERVENTIONS:
Procedure: Positron emission tomography computed tomography (PET/CT) with Intra-hepatic (IAH) injection — Intra-hepatic injection of 68Ga-DOTA-peptides for targeted liver metastases in Positron emission tomography-computed tomography (PET/CT)
Procedure: Positron emission tomography computed tomography (PET/CT) with Intravenous (IV) injection — intravenous injection of 68Ga-DOTA-peptides for targeted liver metastases in Positron emission tomography-computed tomography (PET/CT)
Drug: LUTATHERA® by intra-arterial hepatic (IAH) injection — One treatment dose of LUTATHERA® by IAH injection. The LUTATHERA® by intra-arterial hepatic injection treatment is realised after the conventional treatment by 4 intravenous administrations
Procedure: Scan — Scans after completion of LUTATHERA® treatment injection

SUMMARY:
The management of liver metastases in neuroendocrine neoplasms is challenging. Peptide receptor radionuclide therapy with radiolabeled somatostatin analogs (SSA) is one of the most promising therapeutic options. As liver is the most frequent site of metastatic disease, our project proposes to compare administration of radiolabeled SSA by arterial intrahepatic infusion (experimental approach) vs intravenous administration (conventional). Evaluation will be made by (i) comparing 68Ga-DOTA-peptides uptake after intra-hepatic versus intravenous route (imaging), (ii) by evaluating the safety of an additional intra-hepatic administration of therapeutic radiolabeled SSA (therapy).

DETAILED DESCRIPTION:
Liver metastases of neuroendocrine tumors of gastro-entero-pancreatic origin are one of the most limiting factors of patient survival. Peptide receptor radionuclide therapy with radiolabeled somatostatin analogs (SSA) such as LUTATHERA® represents now a major therapeutic option. As far as these metastases are mainly perfused by the hepatic artery, it could be relevant to deliver the treatment by intra-hepatic route, in order to achieve a maximized dose to the tumour when compared with a systemic conventional administration, while also reducing kidney and bone marrow toxicity. By using radiolabeled SSA for imaging and therapy, the present project aims to compare the uptake of 68Ga-DOTA-peptides after intra-hepatic versus intravenous injections for targeted liver metastases, as well as for dose limiting organs (kidney, spleen, healthy liver, bone marrow) and extra-hepatic lesions if present. The investigators will also evaluate whether the intra-hepatic infusion of one treatment dose of LUTATHERA® after conventional treatment by 4 intravenous administrations, is safe.

Following 4 intravenous administrations of LUTATHERA® in GEP-NET with dominant liver metastases, patients who gave informed consent will be enrolled for 2 PET-scans, the first one after intra-hepatic injection of 68Ga-DOTA-peptides and the second one after intravenous injection for purpose of uptake comparison by 5 liver metastases chosen by radiologists on MRI.

In 10 patients who meet a predefined enhancement ratio of 3, a 5th dose of LUTATHERA® will be administered by intra-arterial hepatic injection. An average enhancement ratio of 3.75 is expected from intra-arterial injection compared to intravenous results. Those 10 patients will be evaluated for 177Lu-DOTA-peptide activity and residence time by SPECT/CT imaging.

Follow-up through 18 months will include clinical examination, MRI and CT scan, as usually performed in these clinical settings and progression

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven well differentiated neuroendocrine tumor (NET) of gastrointestinal or pancreatic origin (GEP).
* Patients are progressive after treatment with cold somatostatin analog (within 12 months according to RECIST), or as soon as the diagnosis is made in case of hepatic invasion > 50% without waiting for tumour progression
* Patient has received 4 standard of care LUTATHERA® cycles
* Liver Metastatic disease dominant or exclusive and assessable by RECIST 1.1, and not amenable to surgical resection after the last cycle
* ECOG performance status 0-2
* Adequate kidney and liver function: creatinine clearance ≥ 50 mL/min, ALT/AST ≤ 2,5x the upper limit of normal
* With no evidence of hematologic alteration after 4 LUTATHERA® cycles: hemoglobin ≥ 8 g/dL, neutrophils ≥ 1500/ mm3, platelets ≥ 75.000/mm3
* Age ≥ 18 years, no superior limit
* Contraception required in pre-menopausal female (Intrauterine device, Progestin Pills, Combined Oral Contraceptives, Monthly Injectables, Progestin Injectables, Combined Patch, Combined Vaginal Ring, Female Sterilization, Vasectomy, Implants) and men for at least 6 months after the last LUTATHERA ® injection.
* Patient´s signed written informed consent
* Patient affiliated to a social security system

Exclusion Criteria:

* Patients with complete response defined by the absence of lesion according to RECIST 1.1 realized during morphological imaging at inclusion (chest-abdomen-pelvis CT scan and hepatic MRI)
* No residual uptake according to standard 177-Lu scintigraphy performed in the clinical routine 24 hours after each LUTATHERA IV treatment
* Carcinoid heart disease (LVEF < 40%)
* Dominant or threatening extrahepatic metastases or that may affect vital prognosis
* Contraindications to intra-hepatic arterial infusion (coagulation disorders, portal thrombosis, intra-hepatic biliary tract dilatation, digestive or biliary anastomosis or fistula, cirrhosis (Child Pugh B8 or C…)
* Serum albumin <30 g/L unless prothrombin time is within the normal range.
* Heart failure, myocardial infarction, stroke, uncontrolled arterial hypertension under optimal treatment (≥ 160/95 mmHg), pulmonary embolism or revascularization procedure, unstable angina pectoris, uncontrolled cardiac arrhythmia, and clinically significant bradycardia during the last 12 months.
* Individuals under legal protection or unable of giving their informed consent
* Pregnancy or breast feeding
* Currently participating to another clinical research protocol
* Individuals under legal protection or unable of giving their informed consent
* MRI scan contraindicated
* LUTATHERA® contraindicated or toxicity during one of the IV administrations leading to a reduction or cancellation of the following dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2027-03-24 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUVmax) on liver metastases | Day 0 (First PET/CT)
  Standardized uptake value (SUVmax) on liver metastase obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on liver metastases | Day 3 (second PET/CT)
  Standardized uptake value (SUVmax) on liver metastase obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides

SECONDARY OUTCOMES:
Standardized uptake value (SUVmax) on healthy liver | Day 0 (First PET/CT)
  Standardized uptake value (SUVmax) on healthy liver obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on healthy liver | Day 3 (second PET/CT)
  Standardized uptake value (SUVmax) on healthy liver obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on kidneys | Day 0 (First PET/CT)
  Standardized uptake value (SUVmax) on kidneys obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on kidneys | Day 3 (second PET/CT)
  Standardized uptake value (SUVmax) on kidneys obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on bone marrow | Day 0 (First PET/CT)
  Standardized uptake value (SUVmax) on bone marrow obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on bone marrow | Day 3 (second PET/CT)
  Standardized uptake value (SUVmax) on bone marrow obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on spleen | Day 0 (First PET/CT)
  Standardized uptake value (SUVmax) on spleen obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on spleen | Day 3 (second PET/CT)
  Standardized uptake value (SUVmax) on spleen obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on associated extra-hepatic metastases | Day 0 (First PET/CT)
  Standardized uptake value (SUVmax) on associated extra-hepatic metastases obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
Standardized uptake value (SUVmax) on associated extra-hepatic metastases | Day 3 (second PET/CT)
  Standardized uptake value (SUVmax) on associated extra-hepatic metastases obtained on PET/CT imaging after injection of 68Ga-DOTA-peptides
177Lu-DOTA-peptide dosimetry | Day 18
  Absorbed dose in different tissue of the 5 hepatic targets, possible extra-hepatic lesions and healthy organs (healthy liver, kidney, bone marrow, spleen)

CONTACTS AND LOCATIONS:
Overall Officials: Ghoufrane TLILI, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Institut Bergonié, Bordeaux
  - Institut de cancérologie du Gard (ICG) - CHU de Nîmes, Nîmes
  - CHU Bordeaux - Hôpital Haut Lévêque, Pessac
  - Institut universitaire du cancer de Toulouse (IUCT) Oncopole, Toulouse